CLINICAL TRIAL: NCT03177317
Title: A Feasibility Study of Reduced Dose of Prophylactic Dexamethasone for Elderly Patients Receiving Moderate Emetogenic Chemotherapies
Brief Title: Reduced Dose of Prophylactic Dexamethasone for Elderly Patients Receiving Moderate Emetogenic Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jin Won Kim, Associate Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1701-379-002
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly patients (>= 70 years of age) (Experimental): Dexamethasone 8mg intravenously before chemotherapy
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8mg IV before chemotherapy on cycle 1 day 1
  Once the complete response is achieved, the dose of dexamethasone will be reduced by 2 mg in the next cycle.

SUMMARY:
Feasibility study to evaluate the efficacy of reduced prophylactic dose of dexamethasone in elderly patients receiving moderate emetogenic chemotherapy

DETAILED DESCRIPTION:
The purpose of this trial is to determine if the dose of dexamethasone used as an antiemetic drug in patients with advanced cancer could be safely reduced.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed colorectal cancer patients with curative resection
* ECOG performance status 0-2
* Provision of signed, written and dated informed consent prior to any study specific procedures
* Receiving adjuvant chemotherapy with FOLFOX (5-FU, leucovorin, oxaliplatin) regimen

Exclusion Criteria:

* Having contraindication to dexamethasone
* Having nausea or vomiting before the start of adjuvant chemotherapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) | 2 weeks
  No emetic episode, no rescue medicine

SECONDARY OUTCOMES:
Complete control (CC) | 2 weeks
  complete response with no more than mild nausea
Complete protection (CP) | 2 weeks
  complete response with no nausea

CONTACTS AND LOCATIONS:
Overall Officials: Jin Won Kim, M.D., PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No